CLINICAL TRIAL: NCT02904057
Title: Evaluation of the Merz Jawline Grading Scale (MJGS) Following Radiesse (+)® Correction of Subcutaneous Volume Loss and Contour Deficits of the Jawline - a Canadian Pilot Study
Brief Title: Evaluation of the MJGS Following Radiesse (+) Injection Into the Jawline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P140891
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2017-06

CONDITIONS: Volume Loss of the Jawline
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment Group (Experimental): The treatment group will receive Radiesse (+) injectable implant up to 3.0 cc per jawline.
  Interventions: Device: Radiesse (+) Injectable Implant
- Control Group (No Intervention): The control group is not treated. They will undergo assessments such as photographs, jaw grading and jaw function tests.

INTERVENTIONS:
Device: Radiesse (+) Injectable Implant — Treated subjects will receive a maximum volume of 3.0 cc of Radiesse (+) per jawline.
  Arms: Treatment Group

SUMMARY:
This study will evaluate the sensitivity of the validated Merz Jawline Grading Scale (MJGS) to detect treatment effects following Radiesse (+) correction of subcutaneous volume loss and contour deficits of the jawline. Treatment effects detected on the MJGS will be correlated with assessments of aesthetic outcomes on the Global Aesthetic Improvement Scale (GAIS) and FACE-Q instrument

DETAILED DESCRIPTION:
A prospective, open label study, in which both right and left jawlines will receive treatment with Radiesse (+). Subjects will be randomized in a 2:1 ratio to either a treatment group or an untreated control group. Jawlines will be assessed by masked evaluators on the MJGS. Treating physicians and treatment group subjects will assess satisfaction on the GAIS. Treatment group subjects will self-report aesthetic outcomes on the FACE-Q instrument.

Treatment subjects will be evaluated at enrollment, and 1, 2 and 4 weeks after enrollment. Control group subjects will be required to be evaluated at enrollment and 4 weeks after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Has right and left jawlines with moderate to severe volume/contour loss as determined by a live, masked evaluator.
2. Is at least 18 years of age.
3. Understands and accepts the obligation not to receive any other procedures below the orbital rim including the neck during participation in the study.
4. Understands and accepts the obligation and is logistically able to present for all scheduled study visits and meet all study requirements.

Exclusion Criteria:

1. Has ever been treated with silicone, PMMA (polymethyl methacrylate), fat injections, poly-L-lactic acid (PLLA; Sculptra®) or permanent dermal fillers below the orbital rim including the neck.
2. Has had surgery on the jawbone or has surgical permanent implant to the face or neck.
3. Has bruxism, masseter muscle hypertrophy or asymmetry of masseter muscles, active temporomandibular joint (TMJ) disease or disorder, or active periodontal disease.
4. Has any medical condition with the potential to interfere with the study or increase the risk of adverse events.
5. Has undergone oral surgery recently or plans to undergo oral surgery procedures during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kuligowski, MD,PHD,MBA, Study Director — Study Director

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 2 sites in Canada.
Pre-assignment Details: A total of 29 participants were screened for the study and all 29 participants were enrolled and treated.
Groups:
- Treatment Group: Radiesse (+) Injectable Implant: Participants received Radiesse+Lidocaine Injectable Implant up to 3.0 cubic centimeter (cc) volume, once within the jawline region of anterior to posterior boundaries (from the mentum to the earlobe) and superior to inferior boundaries (from the lower cheek to the lower body of the jawline).
- Control Group: Untreated: Participants did not receive jawline treatment.
Period: Overall Study
Arm/Group | Treatment Group: Radiesse (+) Injectable Implant | Control Group: Untreated
Started | 19 | 10
Completed | 19 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The randomized set comprised of participants enrolled and randomized into the study.
Groups:
- Treatment Group: Radiesse (+) Injectable Implant: Participants received Radiesse+Lidocaine Injectable Implant up to 3.0cc volume, once within the jawline region of anterior to posterior boundaries (from the mentum to the earlobe) and superior to inferior boundaries (from the lower cheek to the lower body of the jawline).
- Total: Total of all reporting groups
Arm/Group | Treatment Group: Radiesse (+) Injectable Implant | Control Group: Untreated | Total
Number analyzed (Participants) | 19 | 10 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (7.01) | 59.2 (6.39) | 57.3 (6.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 10 | 29
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 19 | 8 | 27
  Black | 0 | 1 | 1
  Other | 0 | 1 | 1
Fitzpatrick skin type [Count of Participants; unit: Participants] — Fitzpatrick skin type depends on the amount of melanin pigment in the skin. This is determined by constitutional colour (white, brown or black skin) and the result of exposure to ultraviolet radiation (tanning). It depends on type of skin where, skin type I:pale or white skin-always burns, does not tan;skin type II:fair skin-burns easily, tans poorly;skin type III:darker white skin-tans after initial burn;skin type IV:light brown skin-burns minimally, tans easily;skin type V:brown skin-rarely burns, tans darkly easily and skin type VI:dark brown or black skin-never burns, always tans darkly.
  Participants
    Type I | 1 | 2 | 3
    Type II | 8 | 4 | 12
    Type III | 10 | 2 | 12
    Type IV | 0 | 0 | 0
    Type V | 0 | 2 | 2
    Type VI | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Jawlines Achieving Greater Than or Equal to (>=) 1-point Improvement on Merz Jawline Grading Scale (MJGS) at Week 4
Description: MJGS is a 5-point scale, where score ranges from (0-4) as, score 0: continuous jawline contour, no downshifting of subcutaneous volume; score 1: mild loss of jawline contour, mild downshifting of subcutaneous volume; score 2: moderate loss of jawline contour, moderate downshifting of subcutaneous volume; score 3: severe loss of jawline contour, severe downshifting of subcutaneous volume and score 4: very severe loss of jawline contour, diffuse mandibular angle, very severe downshifting of subcutaneous volume.
Time Frame: Week 4
Population: The full analysis set (FAS) comprised of the subset of participants in the randomized set for whom the primary efficacy variable was available.
Measure: Number; unit: percentage of jawlines
Units Other Than Participants: Jawlines
Arm/Group | Treatment Group: Radiesse (+) Injectable Implant | Control Group: Untreated
Number analyzed (Participants) | 19 | 10
Number analyzed (Jawlines) | 38 | 20
percentage of jawlines
  Imputed data | 92.1 | 0
  Observed data | 92.1 | 0
Statistical Analysis 1: Comparison: Treatment Group: Radiesse (+) Injectable Implant vs Control Group: Untreated; Imputed Data: Difference between proportion of treatment responders and control responders (P[treatment] - P[control] with confidence interval (CI) was calculated using an exact approach; Test type: Superiority; p < 0.0001, Fisher Exact; Difference between proportion = 92.1, 95% CI 2-sided [73.4 to 98.8]
Statistical Analysis 2: Comparison: Treatment Group: Radiesse (+) Injectable Implant vs Control Group: Untreated; Observed Data: Difference between proportion of treatment responders and control responders (P[treatment] - P[control] with CI was calculated using an exact approach; Test type: Superiority; p < 0.0001, Fisher Exact; Difference between proportion = 92.1, 95% CI 2-sided [73.4 to 98.8]

2. Secondary Outcome: Treatment Group, Radiesse (+) Injectable Implant: Percentage of Jawlines With >=1-point Improvement on the MJGS Versus at Least an Improved Rating on Global Aesthetic Improvement Scale (GAIS) at Week 4
Description: MJGS is a 5-point scale, where score ranges from (0-4) as, score 0: continuous jawline contour, no downshifting of subcutaneous volume; score 1: mild loss of jawline contour, mild downshifting of subcutaneous volume; score 2: moderate loss of jawline contour, moderate downshifting of subcutaneous volume; score 3: severe loss of jawline contour, severe downshifting of subcutaneous volume, and; score 4: very severe loss of jawline contour, diffuse mandibular angle, very severe downshifting of subcutaneous volume. The GAIS is a 7-point scale, where score ranges from (0-7) as: score 0: very much worse; score 1: much worse; score 3: worse; score 4: no change; score 5: improved; score 6: much improved; score 7: very much improved. An "improvement" on the GAIS for the treating investigator was classified as investigators who rated participants as "improved", "much improved", or "very much improved". All other ratings on the GAIS were classified as "no improvement".
Time Frame: Week 4
Population: The FAS comprised the subset of participants in the randomized set for whom the primary efficacy variable was available. The GAIS was assessed only in treated subjects (i.e., not in Control Group: Untreated); therefore, the analysis is on observed cases, where data were available for both assessments.
Measure: Number; unit: percentage of jawlines
Units Other Than Participants: Jawlines
Arm/Group | Treatment Group: Radiesse (+) Injectable Implant
Number analyzed (Participants) | 19
Number analyzed (Jawlines) | 38
percentage of jawlines
  GAIS improvement and MJAS ≥ 1-grade improvement | 92.1
  iGAIS improvement and MJAS no improvement | 7.9
  iGAIS no improvement and MJAS ≥ 1-grade improvement | 0
  iGAIS no improvement and MJAS no improvement | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 4
Description: The investigator asked the participant for adverse events (AEs) systematically at each visit.
Arm/Group | Treatment Group: Radiesse (+) Injectable Implant | Control Group: Untreated
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/10
Other Adverse Events (participants affected / at risk) | 19/19 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group: Radiesse (+) Injectable Implant (N=19) | Control Group: Untreated (N=10)
Injection site bruising (General disorders) | 5 (7) | 0 (0)
Injection site swelling (General disorders) | 12 (23) | 0 (0)
Nodule (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 11 (22) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.